CLINICAL TRIAL: NCT04113083
Title: An Epidemiological Observational Study for Retrospective and Prospective Evaluation of for the Prevalence of Cerebrotendinous Xanthomatosis (CTX) Disease in Neurology and Pediatric Metabolism Clinics in Turkey
Brief Title: An Observational Study for Evaluation of for the Prevalence of Cerebrotendinous Xanthomatosis (CTX) Disease
Acronym: GEN-EYE-II
Status: Terminated | Type: Observational
Why Stopped: Due To Covid-19 there were delays in the arrival of patients to the sites. Due to the rare disease in the study population, no patients who met the inclusion/exclusion criteria were found, and the study was terminated early due to these reasons.
Sponsor: TRPHARM (Industry)
Collaborators: Klinar CRO (Other); Düzen Laboratories Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: TR-CTX-002
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: CTX - Cerebrotendinous Xanthomatosis
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood sampling for cholestanol analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling for cholestanol analysis — Blood sampling will be performed by Düzen Laboratories group for cholestanol

SUMMARY:
The prevalence of CTX in our country is estimated to be 1 / 50.000. The aim of this study is to screen more volunteers by conducting a larger screening from neurology and pediatric metabolism clinics in Turkey.

This observational study was designed retrospectively and prospectively in two stages. In the retrospective section, the patient database and / or patient files will be screened in the neurology and pediatric metabolism clinics and the patients aged 40 and below in the neurology clinics with at least two of the following will be enrolled to the study:

* Ataxia and / or spasticity
* Bilateral cataract (except senile cataract)
* Intellectual limitation
* Non-enhancing hyperintensity on T2 sections in MR imaging of dentate nuclei
* Autosomal recessive transition pattern. (Ex: Relative Marriage)

In the pediatric metabolism centers, cases suspected of CTX and planned to apply the Mignarri Index according to the investigator's opinion will be identified.

ELIGIBILITY:
Inclusion Criteria:

I-1. Giving written informed consent

I-2. Patients in neurology clinics should have been identified with at least two of the following:

* Ataxia and / or spasticity
* Bilateral cataract (except senile cataract)
* Intellectual limitation
* Nonintensitive hyperintensity in T2 sections on MRI of the dentate nucleus
* Forming an autosomal recessive transition pattern. (Ex: Relative Marriage)

I-3. In the pediatric metabolism centers, cases suspected of CTX and planned to apply the Mignarri Index according to the investigator's opinion.

I-4. On the day the patient signed the Informed Consent Form, the patient did not get older than 41 years of age (subjects aged 40 and under will be included in the study)

Exclusion Criteria:

E-1. The patient's ataxia and / or spasticity, cataract, intellectual limitation, and non-contrasted hyperintensity of T2 sections in MR imaging of dentate nuclei with typical MRI findings are due to a known cause other than CTX or other underlying disease.

E-2. The patient has participated in an interventional clinical study in the last 30 days,

E-3. The patient and / or his / her legal representative does not give consent to participate in the study,

E-4. In the opinion of the investigator, the patient is not able to fulfill the working requirements appropriately,

E-5. Pregnancy and / or lactation

E-6. If the patient was 41 years old when included in the study.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 200 patients
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with CTX possibility in Neurology Clinics | 3 years
  - Proportion of patients aged 40 years or younger with at least two of the following (2) in patients with a cholestanol test threshold (3.75 mg / mL) in neurology clinics:
  * Ataxia and / or spasticity
  * Bilateral cataract (except senile cataract)
  * Intellectual limitation
  * Nonintensitive hyperintensity in T2 sections on MRI of the dentate nucleus
  * Forming an autosomal recessive transition pattern. (Ex: Relative Marriage)
Proportion of patients with CTX possibility in Pediatric Metabolism Clinics | 3 years
  - Proportion of cases above the cholestanol test threshold (3.75 mg / mL) in pediatric metabolism centers

SECONDARY OUTCOMES:
Total of Mignarri Suspicion Index (SI) | 3 Years
  Mignarri is a suspicion index, composed of weight-ed scores assigned to indicators such as family history and common systemic and neurological features. The indicators were classified as very strong (score 100), strong (50) or moderate (25). The suspicion index will be applied to study population. Early systemic signs such as catamct, diarrhea and neonatal cholestatic jaundice were considered strong indica- tors, together with neurological features such as intellectual impairment, psychiatric disturbances, ataxia, spastic paraparesis and dentate nuclei abnormalities at MRI. Tendon xanthomas were regarded as very strong indicators, as was an affected sibling. A total score 100 warranted serum cholestanol assessment. Elevated cholestanol or a total score 200, with one very strong or four strong indicators, warranted CYP27Al gene analysis. (Reference: Mignarri et al. J Inherit Metab Dis (2014) 37:421-429)
  -and physical examination results for patients with high cholestanol levels
Cholestanol Levels | 3 Years
  - Cholestanol levels for patients with high cholestanol levels
Patient demographics | 3 Years
  For all screened patients:
  • Demographic data
CTX Family History | 3 Years
  For all screened patients:
  • CTX family history
Presence of consangunious marriage | 3 Years
  For all screened patients:
  • Presence of consanguineous marriage
Frequency of the systemic findings | 3 Years
  For all screened patients:
  • Frequency of the following systemic findings:
  * Tendon xanthomas
  * Chronic diarrhea
  * Prolonged neonatal jaundice
  * Early osteoporosis
Frequency of the neurologic findings | 3 Years
  For all screened patients:
  • Frequency of the following neurological symptoms:
  * Cerebellar ataxia
  * Spastic paraparesis
  * Blateral cataract (except senile cataract)
  * Non-enhancing hyperintensity on T2 sections in MR imaging of dentate nuclei
  * Intellectual disability
  * Psychiatric disorders
  * Epilepsy
  * Parkinson's
  * Polyneuropathy

CONTACTS AND LOCATIONS:
Locations (22):
- Turkey (Türkiye) (22):
  - Çukurova University Medical Faculty Deparment of Metabolism, Adana
  - Çukurova University Medical Faculty Department of Neurology, Adana
  - Ankara Child and Heamatology Hospital Deparment of Metabolism, Ankara
  - Ankara City Hospital, Ankara
  - Ankara Dışkapı Yıldırım Beyazıt Research and Training Hospital Clinic of Neurology, Ankara
  - Gazi University Medical Faculty Department of Pediatric Metabolism, Ankara
  - Hacettepe University Medical Faculty Deparment of Metabolism, Ankara
  - Hacettepe University Medical Faculty Department of Neurology, Ankara
  - Osmangazi University Medical Faculty Department of Neurology, Eskişehir
  - Osmangazi University Medical Faculty Department of Pediatric Metabolism, Eskişehir
  - Bezmi Alem Vakıf University Medical Faculty Department of Neurology, Istanbul
  - Hamidiye Şişli Etfal Research and Training Hospital Clinic of Neurology, Istanbul
  - Hamidiye Şişli Etfal Research and Training Hospital Clinic of Pediatric Metabolism, Istanbul
  - İstanbul University Cerrahpasa Medical Faculty Department of Pediatric Metabolism, Istanbul
  - İstanbul University Cerrahpaşa Medical Faculty Department of Neurology, Istanbul
  - İstanbul University İstanbul Medical Faculty Department of Neurology, Istanbul
  - İstanbul University İstanbul Medical Faculty Department of Pediatric Metabolism, Istanbul
  - Kanuni Sultan Suleyman Research and Training Hospital Clinic of Pediatric Metabolism, Istanbul
  - Medeniyet University Göztepe Research and Training Hospital Clinic of Neurology, Istanbul
  - Mersin City Hospital Department of Metabolism, Mersin
  - Mersin University Medical Faculty Department of Neurology, Mersin
  - Cumhuriyet University Medical Faculty Department of Neurology, Sivas

IPD SHARING:
Plan to Share IPD: No